CLINICAL TRIAL: NCT02012439
Title: The Efficacy and Mechanisms of Cognitive Therapy Compared to Mindfulness-Based Cognitive Therapy in Multiple Sclerosis (MS) Pain
Brief Title: Comparison of the Efficacy and Mechanisms for MBCT and CT for Multiple Sclerosis (MS) Chronic Pain
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Washington (Other)
Collaborators: National Multiple Sclerosis Society (Other)
Responsible Party: Principal Investigator, Dawn Ehde, Professor, Rehabilitation Medicine, University of Washington
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 45416
Record Dates: First submitted 2013-10-22; First posted 2013-12-16 (Estimated); Last update posted 2019-09-16 (Actual); Status verified 2019-09

CONDITIONS: Multiple Sclerosis
Keywords: multiple sclerosis; chronic pain; treatment; nonpharmacological; mindfulness; cognitive therapy
MeSH Terms: conditions — Multiple Sclerosis; Chronic Pain | interventions — Mindfulness-Based Cognitive Therapy; Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Mindfulness Based Cognitive Therapy (Active Comparator): Mindfulness Based Cognitive Therapy
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Cognitive therapy (Active Comparator): Cognitive Therapy
  Interventions: Behavioral: Cognitive Therapy

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: Cognitive Therapy
  Arms: Cognitive therapy

SUMMARY:
Chronic pain is a pervasive, serious problem for many individuals with multiple sclerosis (MS) that is typically inadequately treated by medications alone. There is a critical need to develop and evaluate innovative psychosocial interventions that have the capacity to effectively target the multidimensional nature of MS pain. Cognitive Therapy (CT) is one psychosocial treatment that has been found to be a potentially beneficial treatment for chronic MS pain. This approach teaches patients to identify and replace unhelpful thoughts about pain with helpful, more adaptive thoughts. In addition, over the past decade there has been a steady upsurge of research examining mindfulness meditation-based therapies for the treatment of medical conditions, including symptoms associated with MS. Mindfulness mediation involves training the mind to disengage from automatic thinking patterns to mindfully perceive, in a non-judgmental manner, one's moment-to-moment experiences. This meditation technique teaches patients to become aware of thoughts, emotions, and physical sensations and to recognize that these are transient experiences that can be mindfully perceived, accepted and let go. A promising, more recent trend in treatment development research is the integration of tradition CT with mindfulness-based meditation, an approach referred to as Mindfulness-Based Cognitive Therapy (MBCT). To date, we are the only research group that has adapted and tested a manualized MBCT approach for the treatment of painful medical conditions. Thus, the proposed pilot randomized controlled trial aims to utilize state-of-the-art research methodology to evaluate traditional Cognitive Therapy (CT) compared to an innovative, newly developed Mindfulness-Based Cognitive Therapy (MBCT) protocol for the treatment of chronic pain in individuals with multiple sclerosis. This study will answer three primary questions: (1) Do these treatments work to improve chronic pain for individuals with MS and do these treatment also improve associated symptoms such as depression, fatigue, and engagement in daily activities?; (2) How do these treatments work in individuals with MS, i.e., what factors underlie improvement in outcomes during treatment?; and (3) What are the individual person characteristics that best predict outcome? This will be the first study to examine MBCT within an MS population. The results will lead to the emergence of a novel, much needed additional psychosocial treatment option for patients with chronic MS pain.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of MS obtained by ICD coding list
2. At least 6 months post-diagnosis.
3. At least 18 years old.
4. Read, speak and understand English.
5. Experience chronic pain on a daily basis.
6. Most significant pain problem(s) is or are related to MS.
7. Report an average pain intensity of at least 4 on a 0-10 Numerical Scale in the past week.
8. Most significant pain problem(s) has or have lasted at least six months.
9. Experience ongoing pain with an average intensity of 4 or more on a 0-10 scale when they experience pain.*
10. Have internet access on a daily basis.

Exclusion Criteria:

1. Psychiatric condition or symptoms that would interfere with participation, specifically active suicidal ideation with intent to harm oneself or active delusional or psychotic thinking

-

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-10; Primary Completion 2015-04 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
pain intensity | at post-treatment (5 weeks on average)
  numeric rating scale (0-10 scale)

CONTACTS AND LOCATIONS:
Overall Officials: Dawn Ehde, PhD, Principal Investigator — University of Washington
Locations (1):
- UW Medicine Multiple Sclerosis Center, Seattle, Washington, United States